CLINICAL TRIAL: NCT04660799
Title: A Phase II Comparative, Open-Label, Randomized, Multicenter, China-Only Study to Investigate the Pharmacokinetics, Efficacy and Safety of Subcutaneous Rituximab Versus Intravenous Rituximab Both in Combination With CHOP in Previously Untreated Patients With CD20 Positive Diffuse Large B Cell Lymphoma
Brief Title: A Study on Pharmacokinetics (PK), Efficacy and Safety of Subcutaneous (SC) Versus Intravenous (IV) Rituximab, in Combination With CHOP (Cyclophosphamide, Doxorubicin, Vincristine, Prednisone) in Previously Untreated Participants With CD20 Positive Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO42207
Record Dates: First submitted 2020-11-25; First posted 2020-12-09 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Mabthera, Rituximab, SC, Subcutaneous, DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rituximab IV+CHOP (Active Comparator): Participants will receive 8 cycles of IV rituximab in combination with 6 or 8 cycles of CHOP chemotherapy administered every 3 weeks.
  Interventions: Drug: Rituximab IV; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Paracetamol; Drug: Diphenhydramine hydrochloride or alternative antihistamine
- Rituximab SC+CHOP (Experimental): Participants will receive 1 cycle of IV plus 7 cycles of SC rituximab in combination with 6 or 8 cycles of CHOP chemotherapy administered every 3 weeks.
  Interventions: Drug: Rituximab SC; Drug: Rituximab IV; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Paracetamol; Drug: Diphenhydramine hydrochloride or alternative antihistamine

INTERVENTIONS:
Drug: Rituximab IV — Rituximab will be administered intravenously through Cycle 1-8 at a standard dose of 375 mg/m^2 (milligram per square meter).
  Other Names: MabThera
  Arms: Rituximab IV+CHOP
Drug: Rituximab SC — Rituximab will be administered subcutaneously through Cycle 2-8 at a dose of 1400 milligram (mg).
  Other Names: MabThera
  Arms: Rituximab SC+CHOP
Drug: Rituximab IV — Rituximab will be administered intravenously in Cycle 1 at a standard dose of 375 mg/m^2.
  Other Names: MabThera
  Arms: Rituximab SC+CHOP
Drug: Cyclophosphamide — Cyclophosphamide will be administered IV at a dose of 750 mg/m^2
Drug: Doxorubicin — Doxorubicin will be administered IV at a dose of 50 mg/m^2
Drug: Vincristine — Vincristine will be administered IV at a dose of 1.4 mg/m^2
Drug: Prednisone — Prednisone will be administered orally at a dose of 100 mg/day
Drug: Paracetamol — All participants are required to receive 1000 mg oral paracetamol as premedication prior to starting each infusion of rituximab
Drug: Diphenhydramine hydrochloride or alternative antihistamine — All participants are required to receive 50-100 mg oral diphenhydramine hydrochloride or alternative antihistamine as premedication prior to starting each infusion of rituximab

SUMMARY:
This is a multicenter China-only study to investigate the PK, efficacy and safety of SC rituximab versus IV rituximab, both in combination with CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone) in previously untreated participants with CD20 positive DLBCL. Participants will be randomized to receive eight cycles of rituximab SC or rituximab IV combined with six or eight cycles of standard CHOP chemotherapy. After the end of study treatment, participants will be followed-up every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated CD20 positive diffuse large B-cell lymphoma (DLBCL)
* Participants with an International Prognostic Index (IPI) score of 1 to 5 or IPI score of 0 with bulky disease, defined as one lesion >/=7.5 cm
* At least one bi-dimensionally measurable lesion defined as >/=1.5 cm in its largest dimension on CT scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Left ventricular ejection fraction (LVEF) >/=50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram
* A negative serum pregnancy test or a negative urine pregnancy test within 7 days prior to study treatment
* For men who are not surgically sterile, agreement to use a barrier method of contraception during the treatment period and until >/=12 months after the last dose of rituximab SC or rituximab IV or according to institutional guidelines for CHOP chemotherapy, whichever is longer, and agreement to request that their partners use an additional method of contraception
* For women of reproductive potential who are not surgically sterile, agreement to use adequate methods of contraception during the treatment period and until >/=12 months after the last dose of rituximab SC or rituximab IV or according to institutional guidelines for CHOP chemotherapy, whichever is longer
* Adequate hematologic function confirmed within 14 days prior to randomization

Exclusion Criteria:

* Transformed non-Hodgkin's lymphoma (NHL) or types of NHL other than DLBCL and its subtypes according to World Health Organization classification
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindication to any of the individual components of CHOP, including prior receipt of anthracyclines
* Prior therapy for DLBCL, with the exception of nodal biopsy or local irradiation or surgery for diagnosis
* Prior treatment with cytotoxic drugs or rituximab for another condition (e.g.,rheumatoid arthritis) or prior use of an anti-CD20 antibody
* Current or recent treatment with another investigational drug or participation in another investigational therapeutic study
* Ongoing corticosteroid use (>30 mg/day of prednisone or equivalent)
* Primary CNS lymphoma, blastic variant of mantle cell lymphoma, or histologic evidence of transformation to a Burkitt lymphoma, primary mediastinal DLBCL, primary effusion lymphoma, and primary cutaneous DLBCL
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of significant, uncontrolled concomitant diseases including but not limited to significant cardiovascular disease or pulmonary disease
* Any of the following abnormal laboratory values: creatinine >1.5 upper limit of normal (ULN), aspartate aminotransferase (AST) / alanine aminotransferase (ALT) >2.5ULN, total bilirubin >1.5ULN, prothrombin time - international normalized ratio (PT-INR) / partial thromboplastin time (PTT) / activated partial thromboplastin time (aPTT)>1.5ULN
* Positive test results for chronic hepatitis B (HBV) and or hepatitis C (HCV) infection; Participants with occult or prior HBV infection (defined as negative HBsAg and positive total hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable; Participants positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
* Known history of human immunodeficiency virus (HIV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- China (8):
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Gao Y, Zhang L, Gao S, Yang Y, Zhang Q, Zhang H, He P, Li F, Jing H, Grange S, Bu L, Wang Q, Li L, Huang H. Pharmacokinetics, efficacy, and safety of subcutaneous versus intravenous rituximab in previously untreated Chinese patients with CD20+ diffuse large B-cell lymphoma: a phase II randomized controlled trial. Leuk Lymphoma. 2025 Apr;66(4):680-690. doi: 10.1080/10428194.2024.2439525. Epub 2025 Jan 7. PMID 39773004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 9 centers in China.
Pre-assignment Details: Eligible participants were stratified during randomization according to International Prognostic Index (IPI) scores (IPI 0-2 = low to low-intermediate risk versus IPI 3-5 = high-intermediate to high risk). IPI risk factors include Ann Arbor Stage III or IV, age >60 years, elevated lactate dehydrogenase, Eastern Cooperative Oncology Group (ECOG) performance status >/=2, extranodal involvement >/=2.
Groups:
- Rituximab IV+CHOP: Participants received 8 cycles of intravenous (IV) rituximab in combination with 6 or 8 cycles of CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone) chemotherapy administered every 3 weeks.
- Rituximab SC+CHOP: Participants received 1 cycle of IV plus 7 cycles of subcutaneous (SC) rituximab in combination with 6 or 8 cycles of CHOP chemotherapy administered every 3 weeks.
Period: Overall Study
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Started | 24 | 26
Completed | 17 | 18
Not Completed | 7 | 8
Not completed — Progressive Disease | 1 | 1
Not completed — Death | 2 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.1) | 55.0 (15.5) | 58.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 13 | 17 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 26 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 26 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subcutaneous Serum Rituximab Trough Concentration (Ctrough SC) and Intravenous Serum Rituximab Trough Concentration (Ctrough IV)
Description: For this pharmacokinetics (PK) primary outcome measure the serum rituximab Ctrough for SC and IV administrations were measured at Cycle 7, 21 days after study treatment administration for Cycle 7 (pre-dose of Cycle 8). Geometric mean ratio and 90% confidence interval were estimated based on an ANCOVA model adjusted for tumor load at baseline and are reported in the statistical analysis.
Time Frame: At Cycle 7 (one cycle=21 days), 21 days after study treatment administration, up to 21 weeks
Population: The Per Protocol PK population included all enrolled participants who adhered to the protocol and were assigned to arms as treated. Exclusions were made for the following reasons: missing Ctrough Cycle 7 sample, Cycle 7 Ctrough sample collected with more than 3 days deviation from planned date on Day 22, given a dose that deviated from the planned dose by >20% within 3 cycles (from Cycle 5), a Cycle 7 dose delay of more than 7 days, an assay error impacting Cycle 7 Ctrough measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 19 | 24
micrograms/milliliter (mcg/mL) | 90.7 (21.1) | 137.4 (36.3)
Statistical Analysis 1: Comparison: Rituximab IV+CHOP vs Rituximab SC+CHOP; Geometric mean ratio of Ctrough SC/Ctrough IV and 90% confidence interval were estimated based on an ANCOVA model adjusted for tumor load at baseline; Test type: Non-Inferiority — The lower limit of the two-sided 90% confidence interval (CI) should be above 0.80 in order to show non-inferiority of Ctrough SC versus Ctrough IV; Ratio Ctrough SC/Ctrough IV = 1.52, 90% CI 2-sided [1.28 to 1.79]

2. Secondary Outcome: Observed SC and IV Rituximab Area Under the Curve (AUCsc and AUCiv)
Description: The area under the curve (AUC) for serum rituximab concentration versus time after dosage was measured for SC and IV administrations during Cycle 7. Geometric mean ratio and 90% confidence interval were estimated based on an ANCOVA model adjusted for tumor load at baseline and are reported in the statistical analysis.
Time Frame: During Cycle 7 (one cycle=21 days): pre-dose, within 15 minutes of end of infusion, 24 hours post-dose, Days 3, 7, 15, 21, up to 21 weeks
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 17 | 21
day*mcg/mL | 3050.7 (17.8) | 3806.7 (27.2)
Statistical Analysis 1: Comparison: Rituximab IV+CHOP vs Rituximab SC+CHOP; Geometric mean ratio of AUCsc/AUCiv and 90% confidence interval were estimated based on an ANCOVA model adjusted for tumor load at baseline; Test type: Non-Inferiority — The lower limit of the two-sided 90% confidence interval (CI) should be above 0.80 in order to show non-inferiority of AUCsc versus AUCiv; Geometric mean ratio of AUCsc/AUCiv = 1.25, 90% CI 2-sided [1.10 to 1.42]

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Rituximab
Time Frame: At Cycles 2 and 7 (one cycle=21 days): pre-dose, within 15 minutes of end of infusion, 24 hours post-dose, Days 3, 7, 15, 21, up to 21 weeks
Population: PK analyses were based on all participants with at least one PK assessment. PK analyses were analyzed as treated. Participants were excluded from the PK analysis population if they significantly violated the inclusion or exclusion criteria, deviated significantly from the protocol, or if data were unavailable or incomplete, where the PK analysis might be influenced.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 22 | 26
micrograms per milliliter (mcg/mL)
  Cycle 2 | 200 (18.3) | 144 (29.6)
  Cycle 7: number analyzed (Participants) | 19 | 23
  Cycle 7 | 255 (14.6) | 228 (28.3)

4. Secondary Outcome: Time to Cmax (Tmax) of Rituximab
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: day
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 22 | 26
day
  Cycle 2 | 0.14 [0.09 to 0.94] | 5.42 [1.88 to 13.90]
  Cycle 7: number analyzed (Participants) | 19 | 23
  Cycle 7 | 0.16 [0.10 to 1.03] | 1.99 [1.84 to 6.91]

5. Secondary Outcome: Trough Serum Concentration (Ctrough) of Rituximab
Description: Ctrough was measured at Cycle 2 and Cycle 7, 21 days after study treatment administration for each cycle (pre-dose of Cycle 3 and Cycle 8, respectively).
Time Frame: At Cycles 2 and 7 (one cycle=21 days), 21 days after study treatment administration, up to 21 weeks
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 20 | 26
mcg/mL
  Cycle 2 | 43.2 (26.5) | 63.5 (36.9)
  Cycle 7: number analyzed (Participants) | 17 | 22
  Cycle 7 | 90.7 (21.1) | 137 (36.3)

6. Secondary Outcome: Area Under the Curve (AUC) of Rituximab
Description: AUC is the area under the serum concentration curve over the dosing interval of 21 days during Cycle 2 and Cycle 7.
Time Frame: During Cycles 2 and 7 (one cycle=21 days): pre-dose, within 15 minutes of end of infusion, 24 hours post-dose, Days 3, 7, 15, 21, up to 21 weeks
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 20 | 26
day*mcg/mL
  Cycle 2 | 1730 (21.5) | 2130 (31.1)
  Cycle 7: number analyzed (Participants) | 17 | 21
  Cycle 7 | 3050 (17.8) | 3810 (27.2)

7. Secondary Outcome: Complete Response Rate (CRR) as Determined by the Independent Review Committee (IRC) Using Lugano Response Criteria (LRC) for Malignant Lymphoma
Description: Per LRC, CR based on positron emission tomography- computed tomography (PET-CT) was defined as complete metabolic response (MR) in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass, on 5-point scale (5PS), where, 1= no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. Per LRC, CR based on CT was defined as complete radiologic response in lymph nodes and extralymphatic sites with target nodes/nodal masses regressing to ≤ 1.5 centimeters (cm) in longest transverse diameter (LDi) and no extralymphatic sites of disease; absence of non-measured lesion; organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, immunohistochemistry (IHC) negative.
Time Frame: 6-8 weeks after the last dose of study treatment or 4-8 weeks after last dose of study treatment for early discontinuation (up to approximately 32 weeks)
Population: The intent-to-treat (ITT) population consisted of all randomized participants. Participants are assigned to the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 24 | 26
percentage of participants | 62.5 [40.59 to 81.20] | 80.8 [60.65 to 93.45]
Statistical Analysis 1: Comparison: Rituximab IV+CHOP vs Rituximab SC+CHOP; Stratified by IPI score: IPI 0-2 = low to low-intermediate risk versus IPI 3-5 = high-intermediate to high risk; Test type: Superiority; Difference in CRR = 18.27, 95% CI 2-sided [-8.92 to 45.45]

8. Secondary Outcome: Objective Response Rate (ORR), Complete Response (CR) or Partial Response (PR), as Determined by Investigator and IRC Using Lugano Response Criteria (LRC) for Malignant Lymphoma
Description: ORR=CR+PR. Per LRC: CR by PET-CT: complete MR in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass; no new lesions, no FDG-avid disease in bone marrow; CR by CT: complete radiologic response in lymph nodes and extralymphatic sites with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi, no extralymphatic disease; absence of non-measured lesion; organ enlargement regressing to normal; no new lesions; normal bone marrow; PR by PET-CT: partial MR in lymph nodes and extralymphatic sites with a score of 4 or 5 with reduced uptake compared with baseline + residual masses of any size; no new lesions, residual uptake higher than in normal bone marrow but reduced compared with baseline; PR by CT: ≥ 50% decrease in sum of the product of the perpendicular diameters (SPD) of up to 6 target nodes and extranodal sites; non-measured lesion absent/normal, regressed, but no increase; spleen regressed by >50 % in length beyond normal; no new lesions.
Time Frame: as for outcome 7
Population: The ITT population consisted of all randomized participants. Participants are assigned to the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 24 | 26
percentage of participants
  Investigator | 70.8 [48.91 to 87.38] | 88.5 [69.85 to 97.55]
  IRC | 66.7 [44.68 to 84.37] | 80.8 [60.65 to 93.45]
Statistical Analysis 1: Comparison: Rituximab IV+CHOP vs Rituximab SC+CHOP; Investigator; Stratified by IPI score: IPI 0-2 = low to low-intermediate risk versus IPI 3-5 = high-intermediate to high risk; Test type: Superiority; Difference in ORR Investigator = 17.63, 95% CI 2-sided [-6.86 to 42.11]
Statistical Analysis 2: Comparison: Rituximab IV+CHOP vs Rituximab SC+CHOP; IRC; Stratified by IPI score: IPI 0-2 = low to low-intermediate risk versus IPI 3-5 = high-intermediate to high risk; Test type: Superiority; Difference in ORR IRC = 14.10, 95% CI 2-sided [-12.68 to 40.88]

9. Secondary Outcome: CRR, as Determined by IRC Using International Working Group (IWG) Response Criteria for Non-Hodgkin's Lymphoma (NHL) 1999 Guidelines
Description: CRR was assessed according to the IWG Response Criteria for NHL 1999 guidelines and included CR and CR unconfirmed (CRu). CR was defined as complete disappearance of all clinical and radiographic evidence of disease and disease-related symptoms, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. CRu was defined as disappearance of clinical and radiographic evidence of disease and absence of splenomegaly, with regression of lymph nodes by > 75 % but still >1.5 cm in size, and indeterminate bone marrow assessment.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 24 | 26
percentage of participants | 58.3 [36.64 to 77.89] | 65.4 [44.33 to 82.79]
Statistical Analysis 1: Comparison: Rituximab IV+CHOP vs Rituximab SC+CHOP; Stratified by IPI score: IPI 0-2 = low to low-intermediate risk versus IPI 3-5 = high-intermediate to high risk; Test type: Superiority; Difference in CRR = 7.05, 95% CI 2-sided [-22.49 to 36.59]

10. Secondary Outcome: CRR, as Determined by the Investigator Using Lugano Response Criteria for Malignant Lymphoma
Description: Per LRC, CR based on PET-CT was defined as complete metabolic response (MR) in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass, on 5-point scale (5PS), where, 1= no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of FDG-avid disease in bone marrow. Per LRC, CR based on CT was defined as complete radiologic response in lymph nodes and extralymphatic sites with target nodes/nodal masses regressing to ≤ 1.5 centimeters (cm) in longest transverse diameter (LDi) and no extralymphatic sites of disease; absence of non-measured lesion; organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 24 | 26
percentage of participants | 58.3 [36.64 to 77.89] | 76.9 [56.35 to 91.03]
Statistical Analysis 1: Comparison: Rituximab IV+CHOP vs Rituximab SC+CHOP; Stratified by IPI score: IPI 0-2 = low to low-intermediate risk versus IPI 3-5 = high-intermediate to high risk; Test type: Superiority; Difference in CRR = 18.59, 95% CI 2-sided [-9.55 to 46.73]

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a subject administered a pharmaceutical product, regardless of causal attribution. An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. New disease, exacerbation of existing disease, recurrence of an intermittent medical condition not present at baseline, any deterioration in a laboratory value or other clinical test associated with symptoms or leading to a change in study/concomitant treatment or discontinuation from study drug as well as events related to protocol-mandated interventions are considered AEs. SAEs: any event that met any of these criteria: fatal, life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, medically significant or required intervention to prevent any of the outcomes listed here.
Time Frame: AEs were reported up to 28 days after the last dose (up to approximately 7 months), and SAEs were reported up to 6 months after the last dose of study treatment (up to approximately 1 year)
Population: The safety analysis population consisted of all randomized participants who received at least one dose of study drug, with participants grouped according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 24 | 26
Participants
  AEs | 24 | 26
  SAEs | 11 | 8

12. Secondary Outcome: Number of Participants With Rituximab Administration-related Reactions (ARRs)
Description: Adverse events occurring within 24 hours after administration of rituximab (rituximab IV or rituximab SC) and considered related to the study drug, were considered as ARRs. ARRs could present with one or more of the following symptoms: allergic reaction, arthralgia, bronchospasm, chills, cough, dizziness, dyspnoea, headache, hypertension, hypotension, myalgia, nausea, pruritus, pyrexia, rash, tachycardia, urticaria, vomiting.
Time Frame: Up to 24 hours after the last dose of study treatment (up to approximately 24 weeks)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 24 | 26
Participants | 6 | 7

13. Secondary Outcome: Number of Participants Positive for Anti-drug Antibodies (ADAs) to Rituximab
Description: Reported here is the number of participants who had a positive ADA assay result at baseline or post-baseline. The post-baseline results are divided in treatment-enhanced ADAs and treatment-induced ADAs. Treatment-enhanced ADAs are participants with a positive ADA result at baseline who had one or more post-baseline titer results that was at least 0.60 titer unit greater than the baseline titer result. Treatment-induced ADAs include participants with negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result.
Time Frame: From baseline up to 6 months after the last dose of study treatment (up to approximately 1 year)
Population: The immunogenicity analysis population consisted of all participants with at least one anti-drug antibody (ADA) assessment. Participants were grouped according to treatment received or, if no treatment was received prior to study discontinuation, according to treatment assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
Number analyzed (Participants) | 24 | 26
Participants
  Baseline: number analyzed (Participants) | 23 | 26
  Baseline | 2 | 1
  Post-baseline: Treatment-enhanced | 1 | 0
  Post-baseline: Treatment-induced | 1 | 1

14. Secondary Outcome: Number of Participants Positive for Anti-rHuPH20 Antibodies
Description: Reported here is the number of participants who had a positive anti-rHuPH20 antibody assay result at baseline or post-baseline. The post-baseline results are divided in treatment-enhanced anti-rHuPH20 antibodies and treatment-induced anti-rHuPH20 antibodies. Treatment-enhanced anti-rHuPH20 antibodies are participants with a positive anti-rHuPH20 antibody result at baseline who had one or more post-baseline titer results that was at least 0.60 titer unit greater than the baseline titer result. Treatment-induced anti-rHuPH20 antibodies include participants with negative or missing baseline anti-rHuPH20 antibody result(s) and at least one positive post-baseline anti-rHuPH20 antibody result.
Time Frame: From baseline up to 6 months after the last dose of study treatment (up to approximately 1 year)
Population: The immunogenicity analysis population consisted of all participants with at least one anti-rHuPH20 assessment. Participants were grouped according to treatment received or, if no treatment was received prior to study discontinuation, according to treatment assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab SC+CHOP
Number analyzed (Participants) | 26
Participants
  Baseline | 2
  Post-baseline: Treatment-enhanced | 1
  Post-baseline: Treatment-induced | 1

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (NSAEs) were reported up to 28 days after the last dose (up to approximately 7 months). Serious adverse events (SAEs) and adverse events of special interest (AESIs) were reported up to 6 months after the last dose of study treatment (up to approximately 1 year)
Description: The safety analysis population consisted of all randomized participants who received at least one dose of study drug, with participants grouped according to treatment received.
Arm/Group | Rituximab IV+CHOP | Rituximab SC+CHOP
All-Cause Mortality (participants affected / at risk) | 2/24 | 1/26
Serious Adverse Events (participants affected / at risk) | 11/24 | 8/26
Other Adverse Events (participants affected / at risk) | 24/24 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab IV+CHOP (N=24) | Rituximab SC+CHOP (N=26)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (6) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (7) | 1 (1)
Platelet count decreased (Investigations) | 2 (4) | 0 (0)
White blood cell count decreased (Investigations) | 2 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab IV+CHOP (N=24) | Rituximab SC+CHOP (N=26)
Anaemia (Blood and lymphatic system disorders) | 17 (38) | 25 (60)
Leukocytosis (Blood and lymphatic system disorders) | 4 (12) | 5 (35)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 2 (9)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (10) | 7 (13)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (8)
Fatigue (General disorders) | 2 (5) | 2 (2)
Infusion site reaction (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (9) | 8 (12)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 4 (6) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (7)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 5 (6) | 2 (3)
Lymphocyte count decreased (Investigations) | 11 (34) | 16 (58)
Neutrophil count decreased (Investigations) | 17 (70) | 18 (67)
Neutrophil count increased (Investigations) | 4 (14) | 8 (39)
Platelet count decreased (Investigations) | 14 (39) | 16 (60)
Weight decreased (Investigations) | 6 (6) | 7 (7)
Weight increased (Investigations) | 2 (2) | 2 (2)
White blood cell count decreased (Investigations) | 20 (86) | 21 (91)
White blood cell count increased (Investigations) | 1 (2) | 3 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (10) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (6) | 4 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (16) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (9) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (9) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 10 (10)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 2 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04660799/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04660799/SAP_001.pdf